CLINICAL TRIAL: NCT00564044
Title: Does the Immune Reactivity of Bacteria Cause Vaginal Mesh (Polypropylene) Erosion? - A Ultrastructural, Microbiological and Immunohistochemical Analysis.
Brief Title: The Immune Reactivity of Biofilms in Vaginal Mesh Erosion.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Chang Gung Memorial Hospital (Other)
Collaborators: National Science and Technology Council, Taiwan (Other Government)
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: NMRPD160851; NSC96-2314-B-182-015-MY1; NSC96-2314-B-182-015-MY2
Record Dates: First submitted 2007-11-25; First posted 2007-11-27 (Estimated); Last update posted 2007-11-27 (Estimated); Status verified 2007-08

CONDITIONS: Uterine Prolapse; Urinary Incontinence; Fecal Incontinence
Keywords: biofilm-infection-related immune hyperreactivity; mesh extrusion; mid-urethral sling; determine the immune reactivity of biofilms in mesh erosion
MeSH Terms: conditions — Uterine Prolapse; Urinary Incontinence; Fecal Incontinence

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- 2 (Active Comparator)
  Interventions: Procedure: excision of the protruding mesh and its surrounding vaginal tissue

INTERVENTIONS:
Procedure: excision of the protruding mesh and its surrounding vaginal tissue — A piece of vaginal tissue 12mm*5mm*3mm in sized (for control group) and another piece of vaginal tissue combined with protruding mesh of the same size (for study group) will be obtained respectively for each of the two arms during intervention.

SUMMARY:
Aging, birth trauma and extensive pelvic surgery are the causes known to cause advanced pelvic organ prolaspe, fecal as well as urinary incontinence. Surgical treatment is the last resort to manage the above-mentioned clinical manifestations of pelvic floor disorders except the subject is too frail to receive operation.

In order to improve the outcome of reconstructive pelvic surgery, reinforcement with synthetic mesh or biological material is the modern trend in pelvic repair. Unfortunately no prosthesis including synthetic or biological is ideal because vaginal erosion with mesh extrusion which is the subject of this protocol and other complications were reported continuously. As per the literature, the rate for mesh vaginal extrusion ranged between 2.4 and 17% when polypropylene which is the most popular synthetic material used for the mid-urethral sling or pelvic reconstructive surgery to date. The causes of this complication are still controversial which include rejection, poor quality of tissue, surgical artifact, material of mesh and etc.

A prospective controlled study for the investigation of the cause for mesh vaginal erosion was conducted and the results revealed evidences of immune reactivity after mesh implantation, albeit the evidence was not solid (Am J Obstet Gynecol 2004; 191(6): 1868-1874 ). As per the pilot study initially done by us to determine the biofilm-related-infection, we have found bacterial biofilm could adhere to surfaces and interfaces, i.e. bacteria located in the cells just beneath the contacting surfaces in the electron microscopic (EM) analysis. In addition, soon after bacteria infection, proteins in biofilm undergo conformational changes, making them immunogenic and triggers a typical inflammatory response leading to activation of the complement system. Thus, we plan to use CD (clusters of differentiation) antigens - 4, 8, 20, 25, 40, 68 and quantitative analysis of FoxP3 to determine the function of regulatory T cells in the immune response. In addition, bacterial culture and EM analysis of the excised mesh with surrounding vagina tissue will be performed for further analysis of biofilms.

ELIGIBILITY:
Inclusion Criteria:

* Study arm: Subjects present with mesh erosion in vaginal after placement of polypropylene mesh for either urinary stress incontinence or pelvic organ prolapse.
* Control arm: Subjects present with symptomatic vaginal prolapse but without mesh erosion after placement of polypropylene mesh for either urinary stress incontinence or pelvic organ prolapse.

Exclusion Criteria:

* Study arm: The eligible subjects with fasting sugar level ≥ 180mg/dL, post prandial sugar level ≥ 230mg/dL.
* Control arm: Polypropylene mesh placement less than 6 months.

Ages: 20 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Estimated)
Dates: Start 2007-08; Study Completion 2009-07 (Estimated)

PRIMARY OUTCOMES:
To determine whether bacterial infection with biofilm formation exists in the vaginal tissue with mesh extrusion using bacterial culture and electron microscopic analysis. | 3 years

SECONDARY OUTCOMES:
With the use of immunohistochemical (IHC) analysis of CD 4, 8, 20, 25, 40, 68 and quantitative analysis of Fox P3 (using RT-POR), to determine the function of regulatory T cells in the immune reactivity of biofilms. | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Alex Wang, MD, Principal Investigator — Division of Female Pelvic Medicine and Reconstructive Surgery, Department of OB/GYN, Chang Gung Memorial Hospital; Cheng-Hsun Chiu, MD. PhD, Study Chair — Department of Pediatrics, Chang Gung Memorial Hospital; Yu-Shien Ko, MD, PhD, Study Director — First Cardiovascular Division, Chang Gung Memorial Hospital; Cheng-Tao Lin, MD, Study Director — Division of Gynecological Oncology, Department of OB/GYN, Chang Gung Memorial Hospital; Ren-Chin Wu, MD, Study Director — Department of Surgical Pathology, Chang Gung Memorial Hospital; Tsia-Shu Lo, MD, Study Director — Division of Female Pelvic Medicine and Reconstructive Surgery, Department of OB/GYN, Chang Gung Memorial Hospital; Min-Chi Chen, PhD, Study Director — Biostatistics Center and Department of Public Health, Chang Gung University; Yi-Haou Lin, MD, Study Director — Division of Female Pelvic Medicine and Reconstructive Surgery, Department of OB/GYN, Chang Gung Memorial Hospital
Locations (1):
- Chang Gung Memorial Hospital, Guishan, Taoyuan, Taiwan